CLINICAL TRIAL: NCT02828618
Title: Trial on Radical Upfront Surgery in Advanced Ovarian Cancer
Acronym: TRUST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AGO Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR OP.7/TRUST
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I PDS and chemotherapy (Active Comparator): PDS with maximum effort to achieve the goal of complete gross resection then followed by 6 cycles of standard chemotherapy
  Interventions: Procedure: PDS (Primary Debulkdung Surgery); Procedure: 6 cycles of standard chemotherapy
- Arm II Timing of surgery after 3 cycles of SOC CTX (Experimental): 3 cycles of standard NACT followed by IDS with maximum effort to achieve the goal of complete gross resection followed by 3 more cycles (for a total of 6) of standard chemotherapy
  Interventions: Procedure: Timing of surgery after 3 cycles of standard NACT, IDS; Procedure: IDS; Drug: 3 cycles of standard chemotherapy

INTERVENTIONS:
Procedure: PDS (Primary Debulkdung Surgery) — PDS with maximum effort to achieve the goal of complete gross resection
  Arms: Arm I PDS and chemotherapy
Procedure: 6 cycles of standard chemotherapy — 6 cycles of standard chemotherapy after Primary Debuling Surgery
  Arms: Arm I PDS and chemotherapy
Procedure: Timing of surgery after 3 cycles of standard NACT, IDS — Timing of surgery after 3 cycles of standard NACT
  Arms: Arm II Timing of surgery after 3 cycles of SOC CTX
Procedure: IDS — IDS with maximum effort to achieve the goal of complete gross resection after NACT
  Arms: Arm II Timing of surgery after 3 cycles of SOC CTX
Drug: 3 cycles of standard chemotherapy — 3 more cycles (for a total of 6) of standard chemotherapy after IDS
  Arms: Arm II Timing of surgery after 3 cycles of SOC CTX

SUMMARY:
This study consists of three parts, whereas Part 1 and Part 2 are performed in Germany only, and Part 3 is a multinational trial.

All patients with suspicion of advanced ovarian cancer are detected in the participating study centers in a pre-screening. The study centers will register all patients with suspected ovarian cancer in a screening log. After the patients have given informed consent, they can be enrolled in different parts of the study.

TRUST-Trial: This part compares two strategies in the therapy of advanced ovarian cancer. En detail, this part of the trial will evaluate if one of two strategies of timing surgery within the therapeutic procedures may show any significant advances in terms of overall survival over the other.

DETAILED DESCRIPTION:
Both randomised groups are treated with surgery for complete resection following guideline recommendations and including median laparotomy, complete adhesiolysis, hysterectomy, bilateral salpingo-oophorectomy, omentectomy and (partial) resection of all affected organs (e.g. small or large bowel, peritoneum, spleen, pancreas, peritoneum, urinary tract etc.) as well as pelvic and paraaortic lymphadenectomy if indicated. Patients with significant pleural effusion (>500 mL in the right chest or any pleural effusion in the left chest, assessed either through ultrasound or CT scan) need to undergo video assisted thoracoscopy or open assessment of the pleura prior or during debulking surgery to detect and if possible remove intrathoracic disease.

Group 1: Primary debulking surgery Patients allocated to the primary debulking group undergo surgery followed by 6 cycles of platinum and taxane based chemotherapy.

Recommended systemic treatment Group 1:

It is recommended to start systemic treatment after sufficient regeneration from surgery [45], which will be ideally 2 to 6 weeks (but at the latest 8 weeks) after surgery. The following treatments are recommended:

1. Participation in a prospective randomized trial, as long as participation is possible in case of randomization in either arm of the current study
2. Carboplatin AUC 5-6 / paclitaxel 175 mg/m² q21 / bevacizumab 15mg/KG q21, 6 cycles followed by bevacizumab maintenance therapy for a total of 15 months or until disease progression.
3. Carboplatin AUC 5-6 / paclitaxel 175 mg/m² q21, 6 cycles. Substitution of paclitaxel by docetaxel (75mg/m²) in cases of contraindications to paclitaxel is possible. Maintenance/consolidation therapy inside prospective trials or according to national standard treatments is allowed. Additional treatment outside prospective studies is not recommended.
4. Carboplatin AUC 5 - 6, q21 , 6 cycles in the case of contraindications of combination chemotherapy

Group 2: Interval debulking surgery Patients allocated to the interval debulking surgery group undergo biopsy to confirm ovarian cancer and then 3 cycles of neoadjuvant preoperative platinum and taxane based chemotherapy. Then interval debulking surgery is performed followed by 3 cycles of postoperative platinum and taxane based chemotherapy

Recommended systemic treatment Group 2:

It is recommended to start systemic treatment as soon as possible after biopsy confirmation of ovarian cancer.

The following treatments are recommended for neoadjuvant chemotherapy:

1. Participation in a prospective randomized trial, as long as participation is possible in case of randomization in either arm of the current study
2. Carboplatin AUC5-6 / paclitaxel 175 mg/m² q21, 3 cycles. Substitution of paclitaxel by docetaxel (75mg/m²) in cases of contraindications to paclitaxel is possible.
3. Carboplatin AUC 5-6, q21 , 3 cycles in the case of contraindications of combination chemotherapy

It is recommended to start postoperative chemotherapy after sufficient regeneration from interval debulking surgery, which will be ideally 2 to 6 weeks after surgery. The following treatments are recommended:

1. Participation in a prospective randomized trial, as long as participation is possible in case of randomization in either arm of the current study
2. Carboplatin AUC 5-6 / paclitaxel 175 mg/m² q21 / bevacizumab 15mg/KG q21, 3 cycles followed by bevacizumab maintenance therapy for a total of 15 months or until disease progression.
3. Carboplatin AUC5-6 / paclitaxel 175 mg/m² q21, 3 cycles. Substitution of paclitaxel by docetaxel (75mg/m²) in cases of contraindications to paclitaxel is possible. Maintenance/consolidation therapy inside prospective trials or according to national standard treatments is allowed. Additional treatment outside prospective studies is not recommended.
4. Carboplatin AUC 5-6, q21 , 3 cycles in the case of contraindications of combination chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* suspected or histologically confirmed, newly diagnosed invasive epithelial ovarian cancer FIGO stage IIIB-IV (IV only if resectable metastasis)
* Females aged ≥ 18 years
* Patients who have given their written informed consent
* Good performance status (ECOG 0/1)
* Good ASA score (1/2)
* Preoperative CA 125/CEA ratio ≥ 25 (if CA-125 is elevated)*
* If <25 and/or biopsy with non-serous, non-endometroid histology, esophago-gastro-duodenoscopy (EGD) and colonoscopy mandatory to exclude gastrointestinal primary cancer
* Assessment of an experienced surgeon, that based on all available information, the patient can undergo the procedure and the tumor can potentially be completely resected
* Adequate bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L. This ANC cannot have been induced or supported by granulocyte colony stimulating factors.
* Platelet count ≥ 100 x 109/L.
* Renal function: Serum-Creatinine ≤ 1.5 x institutional upper limit normal (ULN).
* Hepatic function:

  * Bilirubin ≤ 1.5 x ULN.
  * SGOT ≤ 3 x ULN
  * Alkaline phosphatase ≤ 2.5 x ULN.
* Neurologic function: Neuropathy (sensory and motor) less than or equal to CTCAE Grade 1.

Exclusion Criteria:

* Non epithelial ovarian malignancies and borderline tumors
* Secondary invasive neoplasms in the last 5 years (except synchronal endometrial carcinoma FIGO IA G1/2, non melanoma skin cancer, breast cancer T1 N0 M0 G1/2) or with any signs of relapse or activity.
* Recurrent ovarian cancer
* Prior chemotherapy for ovarian cancer or abdominal/pelvic radiotherapy
* Unresectable parenchymal lung metastasis, liver metastasis or bulky lymph-nodes in the mediastinum in CT chest and abdomen/pelvis
* Clinical relevant dysfunctions of blood clotting (including drug induced)
* Any significant medical reasons, age or performance status that will not allow to perform the study procedures (estimation of investigator)
* Pregnancy
* Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent
* Any reasons interfering with regular follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2016-07; Primary Completion 2025-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | Patients will be followed up for a minimum of 5 years after registration/randomisation or until death
  To compare the overall survival (OS) after primary debulking surgery (PDS) versus interval debulking surgery (IDS) following neoadjuvant chemotherapy (NACT) in patients with FIGO (2014) stage IIIB-IVB ovarian, tubal, and peritoneal carcinoma.
  The primary endpoint overall survival time is calculated from the date of randomization until the date of death from any cause or date of last contact (censored observation).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Patients will be followed up for a minimum of 5 years after registration/randomisation or until death
  Progression-free survival time is calculated from the date of randomization until the date of first progressive disease or death, whichever occurs first or date of last contact (censored observation). Progressive disease is defined as clinical or imaging-detected tumor progression or death in cases without prior documented tumor progression.
Progression-free survival 2 (PFS2) | Patients will be followed up for a minimum of 5 years after registration/randomisation or until death
  PFS2 time is calculated from the date of randomization until the date of second progressive disease or death, whichever occurs first or date of last contact (censored observation).
Time to first subsequent anticancer therapy or death (TFST) | Patients will be followed up for a minimum of 5 years after registration/randomisation or until death
  Time to first subsequent anticancer therapy is calculated from the date of randomization until the starting date of the first subsequent anticancer therapy or death, whichever occurs first or date of last contact (censored observation). Maintenance treatments following a cytostatic treatment are not considered separate treatment lines.
Time to second subsequent anticancer therapy or death (TSST) | Patients will be followed up for a minimum of 5 years after registration/randomisation or until death
  Time to second subsequent anticancer therapy is calculated from the date of randomization until the starting date of the second subsequent anticancer therapy or death, whichever occurs first or date of last contact (censored observation). Maintenance treatments following a cytostatic treatment are not considered separate treatment lines.
Quality of life (QoL) | Patients will be followed up for a minimum of 5 years after registration/randomisation or until death
  Quality of life (QoL) as measured by EORTC QLQ-C30 (Version 3), EORTC QLQ-OV28, EQ-5D-3L
Documentation of surgical complications | Patients will be followed up for 1 year after surgery or until death
  Assessment of safety: documentation of surgical complications 28 days after surgery and 1 year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Mahner, Professor MD, Principal Investigator — AGO Study Group
Locations (20):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Medical University of Vienna, Vienna, Austria
- University Hospital, Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Institut Bergonié, Bordeaux
  - Hôpital Européen Georges Pompidou (HEGP), Paris
  - Institute Gustave Roussy, Villejuif
- Germany (8):
  - Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Klinik für Gynäkologie, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Klinik & Poliklinik f. Frauenheilkunde & Geburtshilfe, Dresden
  - Kaiserswerther Diakonie; Florence-Nightingale-Hospital, Düsseldorf
  - Kliniken Essen-Mitte, Evang. Huyssens-Stiftung, Klinik für Gynäkologie und gyn. Onkologie, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Gynäkologie, Hamburg
  - Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Klinikum der Universität München, München
  - Klinikum rechts der Isar, Frauen- und Poliklinik, München
  - Universitätsklinikum Tübingen, Tübingen
- Italy (3):
  - European Institute of Oncology; Gynecologic Cancer Surgery, Milan
  - Fondazione IRCCS Istituto Nazionale Tumori - Milan, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori di Napoli, Naples
- Sweden (2):
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Solna
- Imperial College London, Hammersmith Hospital, Surgery&Cancer, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reuss A, du Bois A, Harter P, Fotopoulou C, Sehouli J, Aletti G, Guyon F, Greggi S, Mosgaard BJ, Reinthaller A, Hilpert F, Schade-Brittinger C, Chi DS, Mahner S. TRUST: Trial of Radical Upfront Surgical Therapy in advanced ovarian cancer (ENGOT ov33/AGO-OVAR OP7). Int J Gynecol Cancer. 2019 Oct;29(8):1327-1331. doi: 10.1136/ijgc-2019-000682. Epub 2019 Aug 15. PMID 31420412